CLINICAL TRIAL: NCT05610722
Title: Use of Insulin Adjustment Device DreaMed Endo Digital During Routine Clinical Use for Subjects With Diabetes Type 1
Acronym: Endo digital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal decision
Sponsor: Rabin Medical Center (Other)
Collaborators: DreaMed Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC057522CTIL
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DreaMed Endo Digital (Other): At each visit, participants who use pump therapy will download their pump and glucose data (V1-V5) as they use to do at clinic visit. Participants who use MDI therapy will use the Endo.Digital App for insulin and glucose documentation and will upload data from their CGM/FGM or glucometer as they use to do at clinic visit.
  In addition, participants will be offered to download data also at home in between study visits, every 3-6 weeks as they feel needed (Phone visits: P1-up to P8). Each time, optimization of pump settings or MDI will be done according to the downloaded data using the Endo.DigitalTM system. The device recommendations for insulin dosing adjustments and diabetes management tips will be reviewed by the treating physician. Each new treatment settings will be approved or edit by the study physician prior to implementation by the participant.
  Interventions: Device: DreaMed Endo Digital

INTERVENTIONS:
Device: DreaMed Endo Digital — The DreaMed Endo.Digital uses information gathered from glucose monitoring (sensor readings or capillary blood glucose measurements), insulin dosing and meal data during daily routine home care. Following a 5-minute data collection and analysis, the algorithm learns and suggests insulin dose adjustments and behavioral tips for optimization of glucose control. The algorithm is designed as an advisory tool for health care professionals.

SUMMARY:
The DreaMed Endo.Digital is indicated for use by healthcare professionals treating individuals with Type 1 Diabetes (T1D) who use insulin pump or multiple daily injections (MDI) as their insulin delivery therapy and monitor their glucose levels by using Continuous Glucose Monitoring (CGM) or Flash Glucose monitoring (FGM), or SMBG above the age of 6 years old and below 30 years.

DreaMed Endo.DigitalTM is indicated for use by healthcare professionals when analyzing CGM/SMBG and pump or MDI data to generate recommendations for optimizing a patient's insulin pump settings for basal rate, carbohydrate ratio (CR), and correction factor (CF); or MDI settings for basal rate, carbohydrate ratio (CR), and correction factor (CF) or Sliding Scale without considering the full clinical status of a particular patient. DreaMed Endo.DigitalTM does not replace clinical judgement.

The proposed study is an open label, interventional study that will include up to 500 participants with type 1 diabetes using insulin pumps or MDI therapy and monitoring glucose levels by continuous glucose monitoring including flash glucose monitoring or SMBG.

The proposed study will be 12 months, therefore will include 5 routine clinic visits.

At each visit, participants who use pump therapy will download their pump and glucose data (V1-V5) as they use to do at clinic visit. Participants who use MDI therapy will use the Endo.Digital App for insulin and glucose documentation and will upload data from their CGM/FGM or glucometer as they use to do at clinic visit.

In addition, participants will be offered to download data also at home in between study visits, every 3-6 weeks as they feel needed (Phone visits). Each time, optimization of pump settings or MDI will be done according to the downloaded data using the Endo.DigitalTM system. The device recommendations for insulin dosing adjustments and diabetes management tips will be reviewed by the treating physician. Each new treatment settings will be approved or edit by the study physician prior to implementation by the participant. At study completion, glycemic control will be evaluated by measured HbA1c and the data obtained from the participant devices and CGM/glucometer metrics, or Endo.Digital App data for MDI users.

ELIGIBILITY:
Inclusion Criteria:

1. Documented T1D for at least 6 months prior to study enrolment
2. Subjects aged 6 years and above and below 30 years
3. HbA1c at inclusion ≤ 10%
4. Subjects using Insulin pump therapy for at least 3 months OR using basal-bolus MDI therapy either carbohydrate counting or using sliding scale for meal bolus:

   1. Basal insulin: Glargine, Degludec, or Detemir and up to sum of 72 units of basal insulin
   2. Bolus insulin: regular insulin, rapid analogues or ultra-rapid analogues
5. Subjects willing to follow study instructions:

   1. For SMBG users: measure capillary blood glucose at least 3 times a day (preferable before each meal). Document blood glucose level, insulin delivery and meals using the App for MDI users and bolus pump calculator for pump users.
   2. For CGM users: Use CGM according to manufacture instructions, document insulin delivery and meals using the App for MDI users and bolus pump calculator for pump users.

Exclusion Criteria:

1. An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.
2. Concomitant diseases/ treatment that influence metabolic control or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety.
3. Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus, such as:

   * Subject has unstable or rapidly progressive renal disease or is receiving dialysis
   * Subject has active proliferative retinopathy
   * Active gastroparesis
4. Participation in any other interventional study
5. Female subject who is pregnant or planning to become pregnant within the planned study duration
6. Subject is in the "honeymoon" phase - i.e. less than 0.5 insulin units/kg per day.
7. Known or suspected allergy to trial products
8. Drug or alcohol abuse.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 month

SECONDARY OUTCOMES:
Percentage of sensor readings below 54 mg/dl | 12 month

OTHER OUTCOMES:
Percentage of sensor readings above 250 mg/dl | 12 month
Percentage of sensor readings 54-70 mg/dl | 12 month
Percentage of sensor readings 180-250mg/dl | 12 month
Mean sensor glucose | 12 month
Glucose variability measured as standard deviation | 12 month
Total insulin dose | 12 month
Total basal insulin dose | 12 month
Total bolus insulin dose | 12 month
Amount of carbohydrates consumed per day | 12 month
Number of recommendations for changes in the treatment plan per patient | 12 month
Number of recommendations for changes in the treatment plan per iteration | 12 month
Number of physician overrides of Endo Digital recommendations | 12 month
Device satisfaction | 12 month
  Device satisfaction evaluate by Healthcare Professionals Post-Intervention Survey
Patient satisfaction from the Mobile App | 12 month
Frequency of home phone visits | 12 month
The time required to review insulin and glucose data, make and send recommendations | 12 month
  The time required to review insulin and glucose data, make and send recommendations will be measured by timer or evaluate by length of visit

CONTACTS AND LOCATIONS:
Overall Officials: Revital Nimri, Dr, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- schneider children medical center of Israel, Petah Tikva, Israel